CLINICAL TRIAL: NCT00992550
Title: Comparison of Hookah and Cigarette Smoking
Acronym: 6114
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10-05144
Record Dates: First submitted 2009-10-06; First posted 2009-10-09 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Smoking
Keywords: hookah; cigarette; smoking
MeSH Terms: conditions — Smoking; Water Pipe Smoking | interventions — Tobacco Products; Smoking Water Pipes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hookah visit, then cigarette visit (Experimental): 4-day inpatient stays for profile of biomarker excretion
  Interventions: Drug: Cigarette; Drug: Hookah
- Cigarette visit, then Hookah visit (Experimental): 4-day inpatient stay for profile of biomarker excretion
  Interventions: Drug: Cigarette; Drug: Hookah

INTERVENTIONS:
Drug: Cigarette
  Other Names: Participant will smoke their usual brand of cigarette
Drug: Hookah
  Other Names: participant will smoke hookah

SUMMARY:
The aim of this study is to compare exposure to tobacco smoke toxins in individuals who smoke both cigarettes and Hookah pipes. Sixteen subjects will be hospitalized on the research ward for two visits of 4 days each. At one visit they will smoke their usual cigarettes in approximately normal frequency, and at the other visit they will smoke Hookah at least twice per day. The order of the visits will be randomized. On the fourth day of each visit (when nicotine, carbon monoxide (CO), and some carcinogen levels will be in a steady state condition), circadian blood and urine and expired air samples will be collected.

DETAILED DESCRIPTION:
Water pipes have been used to smoke various substances for at least four centuries, particularly in certain Asian countries, the Middle East, and Northern Africa. It is estimated that about 100 million people worldwide smoke tobacco in water pipes, which are also known as hookahs (Indian subcontinent and Africa), shisha, borry, goza (Egypt, Saudi Arabia), narghile, argilhe (Jordan, Lebanon, Syria, and Israel), shui yan dai (China), or hubble-bubble.

Water pipes consist of a head (to hold tobacco) which is connected to a body, which in turn is connected to a bowl containing water. A tobacco preparation is placed in the head, and burning charcoal is placed on top of the tobacco, often separated by perforated aluminum foil. The smoker inhales through the mouthpiece, which draws air over the burning charcoal and through the tobacco, creating an aerosol consisting of volatilized and pyrolized tobacco components. The smoke passes through the water in the bowl, cooling the smoke, before being carried through the hose to the smoker.

Hookah tobacco is different from ordinary tobacco in that it is a moist paste-like preparation made from about 30% crude, cut tobacco that is fermented with honey, molasses, and pulp of different fruits to add flavor. Consequently, differences in composition of the products smoked and different temperatures involved in the smoking process result in substantial difference in the composition of hookah smoke compared to cigarette smoke. Hookah smoke is produced at about 450° C compared to about 900° C for cigarettes. In addition, hookah smoke contains charcoal combustion products, which includes substantial amounts of carbon monoxide (3).

In one study, Shihadeh and Saleh found that hookah tobacco produced substantially more tar (100-fold), nicotine (4-fold), carbon monoxide (11-fold), and polycyclic aromatic hydrocarbons (PAHs, 2 to 5-fold) than did comparable amounts of cigarette tobacco. Shafagoj et al compared expired CO and plasma nicotine in cigarette and hookah smokers, and found that the hookah smokers had about 2-fold higher carbon monoxide levels and about 3-fold higher nicotine levels than cigarette smokers. The high delivery of nicotine is unexpected in light of its high water solubility.

Recently, smoking tobacco in water pipes has gained popularity in the US, particularly in areas with sizable Arab-American populations, and also among young non-Arab-Americanpeople, with a number of hookah bars being located near college campuses. A typical session at a hookah bar involves smoking for 45-60 minutes, often with a group of friends (1). In addition, hookahs, hookah tobacco, and accessories are advertised over the Internet. Most users of hookah tobacco believe that it is not addictive, and less harmful than cigarette smoking.

In light of published studies indicating high nicotine and carbon monoxide exposures in hookah smokers, the lack of data on exposure to other toxic substances, and global increases in the prevalence of hookah tobacco use, it is apparent that further research is needed. In the August, 2005 newsletter, Tobacco-Related Disease Research Program (TRDRP) invited research grant applications on all aspects of hookah smoke.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years
* Gender: Equal #s male & female
* Ethnic/Racial Group: Any
* Smoking Status: Smokers of approximately 3 - 10 cigarettes per day; cotinine level of >20 ng/ml.

Exclusion Criteria:

* Medical: Exclude most any chronic illness requiring regular medication.
* Cardiac: History of angina or other serious heart disease; ECG abnormalities on screening.
* Hypertension: screening visit BP of 150/95 or more after 5 min rest
* Respiratory: Asthma - okay if in remission, otherwise exclude.
* Systemic: "Morbidly Obese" Exclude if BMI > 35
* Diabetes: By history
* Chronic Active Hepatitis: By history; elevated liver function tests (LFTs)
* Cancers: By history
* Pregnancy/breastfeeding: By history; positive pregnancy test
* Other tobacco users (pipe, cigar, chewing tobacco, snuff users
* The following list of health conditions are routinely asked at Phone Screening and thus are exclusions "by history":

  * Oral thrush,
  * Glaucoma,
  * Thyroid disease,
  * Urinary retention,
  * Ulcer in past year,
  * Other "life threatening" illness,
  * "Bad veins"; discomfort with blood draws,
  * History of persistent fainting,
  * Psychiatric (Any history of schizophrenia, major depression, or psychiatric hospitalization),
  * Also any condition for which medications are being taken on a regular basis.
* Medications/Supplements: General Exclusion = "any regular oral and/or prescription drug use" with the exception of oral contraceptives and Thyroid (Synthroid)
* Drug/alcohol use: General "no abuse by history", no regular recreational drug use, any intravenous drug abuse (IVDA), recent hx of Tx program No smoking of marijuana or herbal products for one month prior to screening and no smoking of marijuana or herbal products between screening and final study day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
smoke toxin excretion | 10 days

SECONDARY OUTCOMES:
nicotine intake | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital-CTSI CRC, San Francisco, California, United States